CLINICAL TRIAL: NCT07333807
Title: Efficacy of the Pelvic Clock® Device on Functional Recovery After Robotic-Assisted Radical Prostatectomy: A Randomized Controlled Trial
Brief Title: Efficacy of the Pelvic Clock® Device for Functional Recovery After Robotic-Assisted Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, MING-HSIN, YANG, Dr., Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TSGH-B2025051PC
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Radical Prostatectomy
Keywords: prostate cancer; Robotic-assisted radical prostatectomy; Pelvic Clock
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Pelvic Clock Group (Experimental): Participants performed specific exercises using the Pelvic Clock® device in addition to the standard PFMT regimen.
  Interventions: Device: Pelvic Clock®
- Active Comparator: Control Group (Active Comparator): Participants received standard of care with verbal and written instructions for Pelvic Floor Muscle Training (PFMT).
  Interventions: Behavioral: Standard Pelvic Floor Muscle Training (PFMT)

INTERVENTIONS:
Device: Pelvic Clock® — Participants used the device for neuromuscular re-education. Protocol:
  Frequency: 2 sessions per day.
  Duration: 5-10 minutes per session.
  Schedule: Minimum 5 days/week.
  Repetitions: 10-20 repetitions for specific movements (e.g., 12-6 o'clock tilt, 3-9 o'clock tilt). Participants also adhered to the standard PFMT regimen (3-4 sets/day) .
  Arms: Experimental: Pelvic Clock Group
Behavioral: Standard Pelvic Floor Muscle Training (PFMT) — Standard Kegel exercises without assistive devices.
  Frequency: 3-4 sets per day.
  Intensity: Sustain each contraction for 5-10 seconds, followed by 5-10 seconds relaxation.
  Repetitions: 10-15 repetitions per set
  Arms: Active Comparator: Control Group

SUMMARY:
This randomized controlled trial evaluates the efficacy of the Pelvic Clock® device, a proprioceptive neuromuscular facilitation tool, in accelerating functional recovery following Robotic-Assisted Radical Prostatectomy (RARP). The study compares the device intervention against standard Pelvic Floor Muscle Training (PFMT) instructions. The primary goal is to assess the "Trifecta" achievement rate (cancer control, urinary continence, and potency) at 6 months post-surgery.

DETAILED DESCRIPTION:
Functional recovery, specifically urinary continence and erectile potency, remains a major challenge following RARP. Standard PFMT is often limited by poor patient compliance and incorrect muscle isolation. The Pelvic Clock® device is designed to enhance proprioception and facilitate multi-directional control of pelvic floor muscles. Participants undergoing RARP were randomized 1:1 to either the intervention group (Pelvic Clock + Standard PFMT) or the control group (Standard PFMT alone). Functional outcomes, including incontinence (pad weight), erectile function (IIEF-5), and muscle strength (Oxford scale), were assessed at baseline, 1, 3, and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with localized prostate cancer.
* Scheduled for Robotic-Assisted Radical Prostatectomy (RARP).
* Age between 55 and 80 years.

Exclusion Criteria:

* History of neurological disorders affecting pelvic floor function (e.g., -Parkinson's disease, multiple sclerosis, CVA).
* Adjuvant radiotherapy or androgen deprivation therapy.
* Salvage prostatectomy.
* Advanced tumor stage (cT4 or N+).
* Prior pelvic surgery or radiation.
* Cognitive impairment or physical inability to perform prescribed exercises .

Ages: 55 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-12-28 (Actual)

PRIMARY OUTCOMES:
Trifecta Achievement Rate | 6 months post-surgery
  Composite outcome defined as the simultaneous fulfillment of: (1) Cancer control (PSA < 0.2 ng/mL); (2) Urinary continence (0 pads/day); and (3) Potency (ability to achieve erection sufficient for intercourse)

SECONDARY OUTCOMES:
Erectile Function (IIEF-5 Score) | Baseline, 1, 3, and 6 months post-surgery
  Assessed using the International Index of Erectile Function-5. Scores range from 5 to 25, with higher scores indicating better erectile function.
Urinary Incontinence (24-hour Pad Weight) | Baseline, 1, 3, and 6 months post-surgery
  Objective quantification of urinary leakage measured in grams.
Pelvic Floor Muscle Strength (Modified Oxford Scale) | Baseline, 1, 3, and 6 months post-surgery
  Assessed via Digital Rectal Examination (DRE). Scores range from 0 (no contraction) to 5 (strong contraction).
Urinary Quality of Life (EPIC-Urinary Domain) | Baseline, 1, 3, and 6 months post-surgery
  Expanded Prostate Cancer Index Composite - Urinary Domain. Scores range 0-100, higher scores indicate better QoL.
Postoperative Pain (VAS) | Baseline, 1, 3, and 6 months post-surgery
  Visual Analog Scale. Scores range 0-10, lower scores indicate less pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Neihu, Taiwan

IPD SHARING:
Plan to Share IPD: No